CLINICAL TRIAL: NCT00378118
Title: Evaluation of the Use of OraQuick in Children Less Than Eighteen Months Old
Brief Title: Use of OraQuick for Screening HIV in Children Less Than Eighteen Months Old
Status: Completed | Type: Observational
Sponsor: Thrasher Research Fund (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Other Study IDs: ThrasherRF; IRB00001131 of IORG0000774
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: HIV Antibody Testing
Keywords: HIV-1; HIV-2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Abbott-rapid HIV antibody test — Abbott will be used to test serum or whole blood
Other: OraQuick Rapid HIV-1/2 Antibody test — OraQuick for oral fluid HIV antibody testing

SUMMARY:
Blood is the most commonly used specimen to test for HIV. In the past 20 years, use of saliva as an alternative specimen for HIV testing has been explored. Today, very sensitive tests have been formulated and have been used for diagnosing HIV in adults and older children. OraQuick, a rapid test, is one such example. It is a devise that can be used to collect as well test the saliva.

Most studies done on the use of saliva have been carried out in adults and have produced very good results. However very few such studies have been done in children, especially infants. In adults, use of saliva has also highlighted the advantages of ease of collection and increased acceptability of testing.

HYPOTHESIS OraQuick rapid test can detect antiHIV antibodies as well as the Abbott determine test and oral fluid testing is more acceptable than blood testing.

DETAILED DESCRIPTION:
BACKGROUND Serological identification of antibodies to Human Immunodeficiency virus (HIV) in blood is the most widely used method to screen for HIV infection. Use of oral fluid as an alternative to blood sample has been studies the past 20 years and extremely sensitive tests that are able to detect the very low quantities of antibodies found in oral fluid have been formulated and are currently being used. OraQuick rapid test, a combination, collection and testing device that uses both blood and oral fluid was approved for used by the U.S.A, FDA in 2002 and has been tested in adults and older children.

The value of oral fluid in screening for HIV infection in adults is now well established and has been used extensively in field survey and epidemiologic studies. However, these methods have not been studied in children in whom differences in test performance might be expected. Studies in adults have also highlighted the advantages of oral fluid testing, such as ease of collection and high degree of acceptability of testing. This would make oral fluid testing a good alternative for HIV screening in infants, a challenging population in which venipuncture is often difficult or unacceptable.

ELIGIBILITY:
Inclusion Criteria:

* Children aged less than 18 months
* Admission to the Department of Pediatrics for any condition
* Consent from caregiver for HIV testing using both oral fluid and blood r

Exclusion Criteria:

* Age of more than 18 months
* Refusal of consent by caregiver
* Outpatients

Ages: 1 Day to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children admitted to the University Teaching Hospital,Lusaka,Zambia with various illnesses and aged less than 18 months old
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2006-12; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the OraQuick rapid test | one year

SECONDARY OUTCOMES:
Acceptance of HIV testing using oral fluid | one year

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Chunda, Medicine, Principal Investigator — University of Zambia/University Teaching Hospital
Locations (1):
- University Teaching Hospital,Department of Pediatrics, Lusaka, Lusaka Province, Zambia

REFERENCES:
- [Background] Tess BH, Granato C, Parry JV, Santos VA, Lago TG, Newell ML, Dunn DT, Rodrigues LC. Salivary testing for human immunodeficiency virus type 1 infection in children born to infected mothers in Sao Paulo, Brazil. The Sao Paulo Collaborative Study for Vertical Transmission of HIV-1. Pediatr Infect Dis J. 1996 Sep;15(9):787-90. doi: 10.1097/00006454-199609000-00010. PMID 8878222
- See also: This link provides information and guidance on the use of rapid HIV tests — http://www.cdc.gov